CLINICAL TRIAL: NCT06157619
Title: Vitrification of In Vitro Matured Oocytes Following the CAPA-IVM Methodology
Brief Title: Vitrification of Oocytes Matured by CAPA-IVM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centro de Fertilidad y Reproducción Asistida, Peru (Other)
Collaborators: Centro de Estudios e Investigaciones en Biología y Medicina Reproductiva (Unknown)
Responsible Party: Principal Investigator, Sergio Romero, Research Director, Centro de Fertilidad y Reproducción Asistida, Peru
Other Study IDs: SIDISI 23001
Record Dates: First submitted 2023-11-27; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Fertility Preservation
Keywords: In Vitro maturation; Oocyte vitrification; Fertility preservation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 17 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Formulation of Vitrification medium #1: Hydroxypropyl cellulose (HPC), Ethylene glycol, Dimethyl sulfoxide (DMSO) y trehalose
  Interventions: Procedure: Oocyte Vitrification /Warming
- Formulation of Vitrification medium #2: Human serum albumin (HSA), Ethylene glycol, Dimethyl sulfoxide (DMSO) & sucrose
  Interventions: Procedure: Oocyte Vitrification /Warming

INTERVENTIONS:
Procedure: Oocyte Vitrification /Warming — In Vitro matured oocytes will be randomly assigned to any of the two Vitrification protocols

SUMMARY:
It has been reported that the potential of In Vitro matured oocytes might be affected by the vitrification process. In fact, the freezing and thawing procedures routinely used in IVF laboratories, have not yet been adapted to oocytes coming from early antral follicles (normally used for In Vitro Maturation).

This study aims to compare 2 existing protocols for the Vitrification of In Vitro matured oocytes.

DETAILED DESCRIPTION:
This is a single-center non-blinded observational study.

The proposed study will follow a sibling oocyte design in infertile patients. In Vitro Maturation will be performed by using the Capacitation-IVM (CAPA-IVM) methodology.

All cumulus-oocyte complexes (COC) recovered from the patient will be cultured in CAPA medium for 24 hours and then matured for 30 hours (IVM). A minimum of 10 metaphase II (MII) stage oocytes are expected from each CAPA-IVM procedure.

After CAPA-IVM culture, the mature oocytes (MII) will be randomly divided (50/50) into two groups to be subjected to the two vitrification protocols.

In a second step (next cycle), the oocytes from each group will be thawed and fertilized by Intracytoplasmic sperm injection (ICSI). The derived embryos will be cultured to the blastocyst stage (Day 5/6).

The transfer of a single embryo (the one with the best quality) will be carried out. The remaining embryos will be vitrified.

ELIGIBILITY:
Inclusion Criteria:

Either

* Patients with Polycystic ovary morphology: At least 25 follicles (2-9 mm) throughout the ovary and/or increased ovarian volume (>10ml) (it is enough for 1 ovary to meet these criteria)
* Patients with good ovarian reserve: High antral follicle count (AFC): ≥ 20 antral follicles in both ovaries or Anti-müllerian hormone (AMH) value ≥3.5 ng/ml

In both cases, without significant uterine or ovarian anomalies

Exclusion Criteria:

* There are contraindications for the administration of gonadotropins, oral contraceptives and/or other drugs used in the framework of the present study.
* Preimplantation Genetic Testing (PGT) Cycles
* Oocyte donation cycles
* Medical contraindication for pregnancy.
* High grade endometriosis (> grade 2)
* Cases with extremely poor sperm

Ages: 20 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Infertile patients that are subjected to In Vitro maturation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Oocyte survival rate | 6 months
  The survival rate will be calculated by dividing the number of oocytes that survive freezing/thawing by the number of oocytes originally frozen.
  Survival rate will be evaluated per patient, per vitrification protocol.

SECONDARY OUTCOMES:
Oocyte maturation rate | 6 months
  The maturation rate will be calculated by dividing the number of oocytes that mature by the number of oocytes originally plated.
Fertilization rate | 6 months
  The fertilization rate will be calculated by dividing the number of fertilized oocytes by the number of oocytes injected by ICSI.
Cleavage rate | 6 months
  The cleavage rate will be calculated by dividing the number of cleaving embryos by the number of fertilized oocytes.
Rate of Blastocyst formation | 6 months
  The rate of blastocyst formation will be calculated by dividing the number of blastocysts by the number of fertilized oocytes.
Rate of Good quality blastocysts | 6 months
  The rate of good quality blastocysts will be calculated by dividing the number of good quality blastocysts by the number of fertilized oocytes.
Clinical pregnancy rate | 15 months
  The clinical pregnancy rate will be calculated by dividing the number of patients with clinical pregnancy by the number of patients that underwent embryo transfer procedures.
Live birth rate | 15 months
  The live birth rate will be calculated by dividing the number of patients with a live birth by the number of patients that underwent embryo transfer procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Romero, PhD, Principal Investigator — Research Director
Locations (1):
- Centro de Fertilidad y Reproducción Asistida, Lima, Peru

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salama M, Ataman L, Taha T, Azmy O, Braham M, Douik F, Khrouf M, Rodrigues JK, Reis FM, Sanchez F, Romero S, Vega M, Woodruff TK. Building Oncofertility Core Competency in Developing Countries: Experience From Egypt, Tunisia, Brazil, Peru, and Panama. JCO Glob Oncol. 2020 Mar 2;6:360-368. doi: 10.1200/GO.22.00006. eCollection 2020. PMID 35275746
- [Background] Erratum. JCO Glob Oncol. 2022 Mar;8:e2100412. doi: 10.1200/GO.21.00412. No abstract available. PMID 35275733
- [Background] Vuong LN, Le AH, Ho VNA, Pham TD, Sanchez F, Romero S, De Vos M, Ho TM, Gilchrist RB, Smitz J. Live births after oocyte in vitro maturation with a prematuration step in women with polycystic ovary syndrome. J Assist Reprod Genet. 2020 Feb;37(2):347-357. doi: 10.1007/s10815-019-01677-6. Epub 2020 Jan 4. PMID 31902102
- [Background] Sanchez F, Le AH, Ho VNA, Romero S, Van Ranst H, De Vos M, Gilchrist RB, Ho TM, Vuong LN, Smitz J. Biphasic in vitro maturation (CAPA-IVM) specifically improves the developmental capacity of oocytes from small antral follicles. J Assist Reprod Genet. 2019 Oct;36(10):2135-2144. doi: 10.1007/s10815-019-01551-5. Epub 2019 Aug 9. PMID 31399916
- [Background] Braam SC, Ho VNA, Pham TD, Mol BW, van Wely M, Vuong LN. In-vitro maturation versus IVF: a cost-effectiveness analysis. Reprod Biomed Online. 2021 Jan;42(1):143-149. doi: 10.1016/j.rbmo.2020.09.022. Epub 2020 Sep 28. PMID 33132059
- [Background] Coello A, Campos P, Remohi J, Meseguer M, Cobo A. A combination of hydroxypropyl cellulose and trehalose as supplementation for vitrification of human oocytes: a retrospective cohort study. J Assist Reprod Genet. 2016 Mar;33(3):413-421. doi: 10.1007/s10815-015-0633-9. Epub 2016 Jan 11. PMID 26754749
- [Background] Cohen Y, St-Onge-St-Hilaire A, Tannus S, Younes G, Dahan MH, Buckett W, Son WY. Decreased pregnancy and live birth rates after vitrification of in vitro matured oocytes. J Assist Reprod Genet. 2018 Sep;35(9):1683-1689. doi: 10.1007/s10815-018-1216-3. Epub 2018 Jun 4. PMID 29869219